CLINICAL TRIAL: NCT07355790
Title: Evaluation of the Comfort Increase Provided by an Additional Foam Pad on a Lumbar Belt "Cellacare Lumbal Classic - Lohmann & Rauscher" and Its Biophysical Impact
Brief Title: Evaluation of the Comfort Increase Provided by an Additional Foam Pad on a Lumbar Belt and Its Biophysical Impact
Acronym: CONFORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Lohmann & Rauscher (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25CH171; ANSM (Other: 2025-A01675-44)
Record Dates: First submitted 2025-11-27; First posted 2026-01-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain; Healthy Volunteer
Keywords: Lumbar belt; back insert; confort
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group with additional back insert of a lumbar belt (Experimental): Additional back insert of a lumbar belt
  Interventions: Device: MRI evening 1
- Control group with lumbar belt (Active Comparator): a lumbar belt
  Interventions: Device: MRI evening 2
- Control group without lumbar belt (Sham Comparator): without lumbar belt
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI in the evening without lumbar belt
  Arms: Control group without lumbar belt
Device: MRI evening 2 — MRI in the evening after wearing the lumbar belt for one day
  Arms: Control group with lumbar belt
Device: MRI evening 1 — MRI in the evening after wearing the lumbar belt with additional back insert for one day
  Arms: Experimental group with additional back insert of a lumbar belt

SUMMARY:
The spine is the central musculoskeletal system of the back. It carries and supports a major part of the body weight and ensures simultaneously the trunk's mobility, particularly the mobility of the lumbar spine and the head's mobility by moving the cervical spine. Back pain in the lumbar spine area is the most common kind of pain with a prevalence of 60 to 70 per cent in industrialized countries (Jellema2001).

DETAILED DESCRIPTION:
Back orthosis permits temporary support and stress reduction (in terms of load) of the concerned structures and first of all intervertebral disks. The aim of this study is to evaluate the comfort variation with and without the additional back insert, with the hypothesis that a more comfortable lumbar belt would improve the care observance. This study also aims to verify the relevancy of objective indicators such as pressure measurement and disk hydration for the added benefice of the back insert.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, men or women, aged 18 to 50 years old without lumbar pathology.
* Volunteer beneficiary of a social security scheme.
* Volunteer informed about the study and having co-signed a consent form to participate to the study with the investigator

Exclusion Criteria:

* Protected persons
* Pregnant or breastfeeding women
* Persons deprived of freedom, hospitalised without consent, hospitalised with other ends then research.
* Adults under legal protection (protection of vulnerable adults) or not able to express consent.
* Persons showing gait difficulties (test on treadmill) or with neurological/joint pathologies promoting falls (Parkinson, hemiplegia, …)
* Patient seen by a doctor for lumbar pain in the 2 months prior to the inclusion.
* Patient suffering from scoliosis
* Refusal of consent
* Contraindication to MRI
* Patient carrying an internal electronic device (pacemaker, neurostimulator, insulin pump…)
* Patient with known allergies to one of the product components (e.g. latex)
* During the first MRI, volunteers showing prior signs of lower back pain or discopathy will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Comfort | Day1
  Comfort is measuring with a scale : 0 = uncomfortable, 10 = extremely comfortable

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France